CLINICAL TRIAL: NCT04931199
Title: A Mobile Health Solution to Improve Between-Session Skills Practice in Youth Mental Health Treatment
Brief Title: A Mobile Health Solution for Homework During CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 002313; K23MH118482 (NIH)
Record Dates: First submitted 2021-06-02; First posted 2021-06-18 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Anxiety; Depression; Posttraumatic Stress Disorder
Keywords: mhealth; mental health; youth mental health; adolescent mental health; homework
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic; Psychological Well-Being | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- CBT+App (Experimental)
  Interventions: Behavioral: CBT+App

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — The standard of care procedures for children with clinically elevated anxiety, depression, and PTSD is traditional CBT from their mental health provider.
  Arms: CBT
Behavioral: CBT+App — Participants receive CBT as usual enhanced with a simple, HIPAA compliant, web-based application to help mental health providers implement homework during CBT with children with elevated PTSD, anxiety, and/or depression, and their caregivers. The three major components of the app help providers to (1) Practice interactive, digitized CBT exercises with patients in-session; (2) Remind patients to practice CBT exercises for homework, and (3) Review homework during the next session.
  Arms: CBT+App

SUMMARY:
The purpose of this study is to preliminarily evaluate a web-based app to improve provider implementation and patient engagement in homework (i.e., between-session practice of skills learned during therapy) during child mental health treatment by conducting a small-scale feasibility trial in community practice settings comparing Cognitive Behavioral Therapy (CBT) to CBT enhanced with the app.

ELIGIBILITY:
Inclusion Criteria:

Providers:

* English-speaking
* Mental health providers who have obtained at least a master's degree in social work, counseling, clinical psychology, or related field
* Carry active child mental health treatment caseloads
* Have a laptop, tablet, or smartphone with internet access

Youth:

* English-speaking
* Youth Ages 7-17 years
* Clinically elevated anxiety and depression as indicated by a T-score ≥ 65 on the Revised Children's Anxiety and Depression Scale-25 Child Version (RCADS-25-Y) and/or Revised Children's Anxiety and Depression Scale-25 Parent Version (RCADS-25-P) or total score ≥ 15 on the Child and Adolescent Trauma Screen - Youth Report (CATS-Y) and/or Child and Adolescent Trauma Screen - Caregiver Report (CATS-P)
* Have a laptop, tablet, or smartphone with internet access

Caregivers:

* English-speaking
* Adult (≥18 years old)
* Caregivers of a youth who meets eligibility criteria
* Have internet and smartphone access.

Exclusion Criteria:

Youth with self- or caregiver-reported:

* Active psychotic symptoms (e.g., hallucinations, delusions)
* Significant cognitive disability, developmental delays, or pervasive developmental disorder.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Revised Children's Anxiety and Depression Scale-25 Child Version (RCADS-25-Y) | Baseline
  The Revised Children's Anxiety and Depression Scale-25 Child Version (RCADS-25-Y) is a 25-item self-report questionnaire that assesses levels of anxiety and depression in youth. Total, Total Anxiety, and Total Depression T-scores range from 0 to >80 with higher scores reflecting greater symptom severity.
Revised Children's Anxiety and Depression Scale-25 Child Version (RCADS-25-Y) | 3-Months Post-Baseline
  The Revised Children's Anxiety and Depression Scale-25 Child Version (RCADS-25-Y) is a 25-item self-report questionnaire that assesses levels of anxiety and depression in youth. Total, Total Anxiety, and Total Depression T-scores range from 0 to >80 with higher scores reflecting greater symptom severity.
Revised Children's Anxiety and Depression Scale-25 Child Version (RCADS-25-Y) | 6-Months Post-Baseline
  The Revised Children's Anxiety and Depression Scale-25 Child Version (RCADS-25-Y) is a 25-item self-report questionnaire that assesses levels of anxiety and depression in youth. Total, Total Anxiety, and Total Depression T-scores range from 0 to >80 with higher scores reflecting greater symptom severity.
Revised Children's Anxiety and Depression Scale-25 Parent Version (RCADS-25-P) | Baseline
  The Revised Children's Anxiety and Depression Scale-25 Parent Version (RCADS-25-P) is a 25-item caregiver-report questionnaire that assesses levels of anxiety and depression in youth. Total, Total Anxiety, and Total Depression T-scores range from 0 to >80 with higher scores reflecting greater symptom severity.
Revised Children's Anxiety and Depression Scale-25 Parent Version (RCADS-25-P) | 3-Months Post-Baseline
  The Revised Children's Anxiety and Depression Scale-25 Parent Version (RCADS-25-P) is a 25-item caregiver-report questionnaire that assesses levels of anxiety and depression in youth. Total, Total Anxiety, and Total Depression T-scores range from 0 to >80 with higher scores reflecting greater symptom severity.
Revised Children's Anxiety and Depression Scale-25 Parent Version (RCADS-25-P) | 6-Months Post-Baseline
  The Revised Children's Anxiety and Depression Scale-25 Parent Version (RCADS-25-P) is a 25-item caregiver-report questionnaire that assesses levels of anxiety and depression in youth. Total, Total Anxiety, and Total Depression T-scores range from 0 to >80 with higher scores reflecting greater symptom severity.
Child and Adolescent Trauma Screen - Youth Report (CATS-Y) | Baseline
  The Child and Adolescent Trauma Screen - Youth Report (CATS-Y) is a 25-item self-report questionnaire that assesses levels of post traumatic distress in youth. Total scores range from 0 to 60 with higher scores reflecting greater symptom severity.
Child and Adolescent Trauma Screen - Youth Report (CATS-Y) | 3-Months Post-Baseline
  The Child and Adolescent Trauma Screen - Youth Report (CATS-Y) is a 25-item self-report questionnaire that assesses levels of post traumatic distress in youth. Total scores range from 0 to 60 with higher scores reflecting greater symptom severity.
Child and Adolescent Trauma Screen - Youth Report (CATS-Y) | 6-Months Post-Baseline
  The Child and Adolescent Trauma Screen - Youth Report (CATS-Y) is a 25-item self-report questionnaire that assesses levels of post traumatic distress in youth. Total scores range from 0 to 60 with higher scores reflecting greater symptom severity.
Child and Adolescent Trauma Screen - Caregiver Report (CATS-P) | Baseline
  The Child and Adolescent Trauma Screen - Caregiver Report (CATS-P) is a 25-item caregiver-report questionnaire that assesses levels of post traumatic distress in youth. Total scores range from 0 to 60 with higher scores reflecting greater symptom severity.
Child and Adolescent Trauma Screen - Caregiver Report (CATS-P) | 3-Months Post-Baseline
  The Child and Adolescent Trauma Screen - Caregiver Report (CATS-P) is a 25-item caregiver-report questionnaire that assesses levels of post traumatic distress in youth. Total scores range from 0 to 60 with higher scores reflecting greater symptom severity.
Child and Adolescent Trauma Screen - Caregiver Report (CATS-P) | 6-Months Post-Baseline
  The Child and Adolescent Trauma Screen - Caregiver Report (CATS-P) is a 25-item caregiver-report questionnaire that assesses levels of post traumatic distress in youth. Total scores range from 0 to 60 with higher scores reflecting greater symptom severity.

SECONDARY OUTCOMES:
Homework Rating Scale II (HRS II) | Weekly between Baseline and 3-Months Post-Baseline
  The Homework Rating Scale II (HRS II) is a 4-item self-report questionnaire that assesses levels of homework adherence in cognitive behavior therapy. Total scores range from 0 to 8 with higher scores reflecting greater homework adherence.
Homework Adherence and Competence Scale (HAACS) | Weekly between Baseline and 3-Months Post-Baseline
  The Homework Adherence and Competence Scale (HAACS) is a 19-item independent evaluator-rated instrument that assesses therapists' adherence and competence in reviewing, designing, and assigning homework assignments in cognitive behavior therapy. Total scores range from 0 to 30 for Reviewing homework, 0 to 54 for Designing homework, and 0 to 30 for Assigning homework, with higher scores reflecting greater adherence/competence.
Child and Adolescent Disruptive Behavior Inventory (CADBI) | Baseline
  The Child and Adolescent Disruptive Behavior Inventory (CADBI) is a 25-item caregiver-report questionnaire that assesses levels of post traumatic distress in youth. Total scores range from 0 to 200 with higher scores reflecting greater symptom severity.
Child and Adolescent Disruptive Behavior Inventory (CADBI) | 3-Months Post-Baseline
  The Child and Adolescent Disruptive Behavior Inventory (CADBI) is a 25-item caregiver-report questionnaire that assesses levels of post traumatic distress in youth. Total scores range from 0 to 200 with higher scores reflecting greater symptom severity.
Child and Adolescent Disruptive Behavior Inventory (CADBI) | 6-Months Post-Baseline
  The Child and Adolescent Disruptive Behavior Inventory (CADBI) is a 25-item caregiver-report questionnaire that assesses levels of post traumatic distress in youth. Total scores range from 0 to 200 with higher scores reflecting greater symptom severity.
KIDSCREEN-10 Index Child and Adolescent Version (KIDSCREEN-10-Y) | Baseline
  The KIDSCREEN-10 Index Child and Adolescent Version (KIDSCREEN-10-Y is a 10-item self-report questionnaire that assesses levels of quality of life in youth. Total T-scores range from 0 to >80 with higher scores reflecting greater quality of life.
KIDSCREEN-10 Index Child and Adolescent Version (KIDSCREEN-10-Y) | 3-Months Post-Baseline
  The KIDSCREEN-10 Index Child and Adolescent Version (KIDSCREEN-10-Y is a 10-item self-report questionnaire that assesses levels of quality of life in youth. Total T-scores range from 0 to >80 with higher scores reflecting greater quality of life.
KIDSCREEN-10 Index Child and Adolescent Version (KIDSCREEN-10-Y) | 6-Months Post-Baseline
  The KIDSCREEN-10 Index Child and Adolescent Version (KIDSCREEN-10-Y is a 10-item self-report questionnaire that assesses levels of quality of life in youth. Total T-scores range from 0 to >80 with higher scores reflecting greater quality of life.
KIDSCREEN-10 Index Parent Version (KIDSCREEN-10-P) | Baseline
  The KIDSCREEN-10 Index Parent Version (KIDSCREEN-10-P) is a 10-item caregiver-report questionnaire that assesses levels of quality of life in youth. Total T-scores range from 0 to >80 with higher scores reflecting greater quality of life.
KIDSCREEN-10 Index Parent Version (KIDSCREEN-10-P) | 3-Months Post-Baseline
  The KIDSCREEN-10 Index Parent Version (KIDSCREEN-10-P) is a 10-item caregiver-report questionnaire that assesses levels of quality of life in youth. Total T-scores range from 0 to >80 with higher scores reflecting greater quality of life.
KIDSCREEN-10 Index Parent Version (KIDSCREEN-10-P) | 6-Months Post-Baseline
  The KIDSCREEN-10 Index Parent Version (KIDSCREEN-10-P) is a 10-item caregiver-report questionnaire that assesses levels of quality of life in youth. Total T-scores range from 0 to >80 with higher scores reflecting greater quality of life.
Generalized Anxiety Disorder-7 (GAD-7) | Baseline
  The Generalized Anxiety Disorder scale-7 (GAD-7) is a seven-item diagnostic tool validated in both the primary care setting and the general population
Generalized Anxiety Disorder-7 (GAD-7) | 3-Months Post-Baseline
  The Generalized Anxiety Disorder scale-7 (GAD-7) is a seven-item diagnostic tool validated in both the primary care setting and the general population
Generalized Anxiety Disorder-7 (GAD-7) | 6-Months Post-Baseline
  The Generalized Anxiety Disorder scale-7 (GAD-7) is a seven-item diagnostic tool validated in both the primary care setting and the general population
Patient Health Questionnaire-8 (PHQ-8) | Baseline
  The eight-item Patient Health Questionnaire depression scale (PHQ-8) is established as a valid diagnostic and severity measure for depressive disorders in large clinical studies
Patient Health Questionnaire-8 (PHQ-8) | 3-Months Post-Baseline
  The eight-item Patient Health Questionnaire depression scale (PHQ-8) is established as a valid diagnostic and severity measure for depressive disorders in large clinical studies
Patient Health Questionnaire-8 (PHQ-8) | 6-Months Post-Baseline
  The eight-item Patient Health Questionnaire depression scale (PHQ-8) is established as a valid diagnostic and severity measure for depressive disorders in large clinical studies
Working Alliance Inventory - Short Revised - Client Version (WAI-SR) | 3-Months Post-Baseline
  The Working Alliance Inventory-Short Revised (WAI-SR) is a 12-item measure for the assessment of the therapeutic alliance.
Child/Adolescent Satisfaction Questionnaire (CASQ-Y) | 3-Months Post-Baseline
  CASQ is a 14 item questionnaire administered to children and youth involved with mental health services. It is identical to the parent version and measures three dimensions of satisfaction with mental health services:
Caregiver Satisfaction Questionnaire (CSQ-P) | 3-Months Post-Baseline
  Client Satisfaction Questionnaire (CSQ-8) examines the level of consumer satisfaction with children's (ages 8 to 17 years) outpatient mental health services
Attitudes Toward Homework Questionnaire (ATHQ) | Baseline
  A self-report assessing practitioners' demographic characteristics, use of homework assignments and attitudes towards the use of homework assignments in psychotherapy
Attitudes Toward Homework Questionnaire (ATHQ) | 3-Months Post-Baseline
  A self-report assessing practitioners' demographic characteristics, use of homework assignments and attitudes towards the use of homework assignments in psychotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT04931199/Prot_SAP_000.pdf